CLINICAL TRIAL: NCT01075386
Title: Expression and Function of Ghrelin and Its Receptor, Growth Hormone Secretagogue Receptor TWEAK Protein and Its Receptor Fn14 in Human Endometrial Cancer
Brief Title: The Effects of the Endocrine System on Endometrial Cancer
Acronym: Ghrelin
Status: Completed | Type: Observational
Sponsor: Queensland Centre for Gynaecological Cancer (Other Government)
Collaborators: Greenslopes Private Hospital (Unknown); The University of Queensland (Other); Sullivan Nicolaides Pathology (Industry)
Responsible Party: Sponsor
Other Study IDs: Endo01
Record Dates: First submitted 2010-02-23; First posted 2010-02-25 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Endometrial Cancer
Keywords: Hysterectomy; Endometrial cancer; Benign; Endocrine system; Tissue collection
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Endometrial tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Grade 2: Patients with Endometrial cancer of Grade 1 differentiation
- Benign: Patients without endometrial cancer
- Grade 1: Patients with Endometrial cancer of Grade 2 differentiation
- Grade 3: Patients with Endometrial cancer of Grade 3 differentiation

SUMMARY:
Endometrial cancer usually begins in the endometrium, which is the tissue lining of the uterus. Endometrial cancer is the most commonly diagnosed gynaecological malignancy in Australia. It affects 1 in 80 Australian women and there are about 1400 new cases and 260 deaths from the disease every year. Most affected women are aged between 50 and 70 years. The purpose of this study is to investigate the possible role of the endocrine system in the regulation of human endometrial cancer. By looking at the laboratory results of people with endometrial cancer and also those without endometrial cancer we hope to gain a better understanding of how endometrial cancer develops and progresses. This may lead to the development of new, effective therapies for endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

* women aged 18 years or older
* having a hysterectomy for the treatment of endometrial cancer, fibroids, chronic pelvic pain or abnormal uterine bleeding
* have provided informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with endometrial cancer and patients who are having a hysterectomy for non-cancerous conditions such as fibroids, chronic pelvis pain or abnormal uterine bleeding are eligible for the study
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2011-08 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chen Chen, MD PhD, Study Chair — The University of Queensland
Locations (1):
- Greenslopes Private Hospital, Greenslopes, Queensland, Australia